CLINICAL TRIAL: NCT02289339
Title: Experience With Percutaneous Transcatheter Aortic Valve Implantation in Patients With Symptomatic Aortic Valve Disease in Two German Centers
Brief Title: Everyday Practice With Transcatheter Aortic Valve Implantation
Acronym: EVERY-TAVI
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Julinda Mehilli, Prof. MD, LMU Klinikum
Other Study IDs: MucS001-14
Record Dates: First submitted 2014-11-08; First posted 2014-11-13 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAVI patients: all patients undergoing transcatheter aortic valve prostheses implantation
  Interventions: Device: aortic valve prostheses

INTERVENTIONS:
Device: aortic valve prostheses — balloon-expandable and self-expandable aortic valve prostheses
  Other Names: CoreValve, CoreValveE, Sapien XT, Sapien S3, Lotus

SUMMARY:
The purpose of this registry is to document the everyday practice in our centers with minimal invasive treatment of patients with aortic valve disease who were considered suitable for transfemoral aortic valve implantation by heart team.

DETAILED DESCRIPTION:
The TAVI program in our center started on November 2007. As part of the national policy for quality assurance in medicine a detailed clinical characterization of the TAVI-population was required. Furthermore, a detailed description of the procedure and peri-procedural complications until discharge was required. In our center we designed and are routinely using a TAVI database which fulfills the authority requirements as well as has additional data needed for planning and documentation of TAVI procedure. Since there is already a considerable number of TAVI patients in this database we aim to perform statistical analyses answering different question in this filed.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis
* Intermediate-to-high risk for surgery
* Heart team decision

Exclusion Criteria:

* Contraindication to transfemoral TAVI procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with aortic valve stenosis suitable for transfemoral transcatheter aortic valve implanation
Sampling Method: Non-Probability Sample
Enrollment: 2370 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-20 (Actual)

PRIMARY OUTCOMES:
incidence of post-TAVI aortic regurgitation | 30 days
  echocardiographicall and angiographycally determined

SECONDARY OUTCOMES:
incidence of bleeding complications | 30 days
  defined according to BARC and VARC-2 classification
mortality | 30 days
  all-cause and cardio/cerebrovascular death
mortality rate | 2-years
  all-cause and cardio/cerebrovascular death
mortality rate | 5-years
  all-cause and cardio/cerebrovascular death
incidence of cerebrovascular events | 30 days
  stroke or TIA
incidence of cerebrovascular events | 2-years
  stroke or TIA
incidence of cerebrovascular events | 5-years
  stroke or TIA
incidence of new pacemaker implantation | 30-day
  pacemaker after TAVI
incidence of new pacemaker implantation | 1-year
  pacemaker after TAVI

OTHER OUTCOMES:
incidence of vascular complications | 30 days
  defined according to VARC-2 classification
incidence of re-hospitalisation | 2-year
  new unplanned hospital stay due to cardiovascular und cerebrovascular reasons
incidence of re-hospitalisation | 5-year
  new unplanned hospital stay due to cardiovascular und cerebrovascular reasons

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, Prof. MD, Principal Investigator — Cardiology Department, Munich University Clinic, Ludwig-Maximilian University; Steffen Massberg, Prof. MD, Study Chair — Cardiology Department, Munich University Clinic, Ludwig-Maximilian University
Locations (2):
- Germany (2):
  - Cardiology Department, Segeberger Kliniken, Bad Segeberg
  - Department of Cardiology, Munich University Clinic, Ludwig-Maximilian University, Munich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jochheim D, Zadrozny M, Ricard I, Sadry TM, Theiss H, Baquet M, Schwarz F, Bauer A, Khandoga A, Sadoni S, Pichlmaier M, Hausleiter J, Hagl C, Massberg S, Mehilli J. Predictors of cerebrovascular events at mid-term after transcatheter aortic valve implantation - Results from EVERY-TAVI registry. Int J Cardiol. 2017 Oct 1;244:106-111. doi: 10.1016/j.ijcard.2017.03.003. PMID 28784441
- [Result] Mehilli J, Jochheim D, Abdel-Wahab M, Rizas KD, Theiss H, Spenkuch N, Zadrozny M, Baquet M, El-Mawardy M, Sato T, Lange P, Kuppatt C, Greif M, Hausleiter J, Bauer A, Schwarz F, Pichlmaier M, Hagl C, Richardt G, Massberg S. One-year outcomes with two suture-mediated closure devices to achieve access-site haemostasis following transfemoral transcatheter aortic valve implantation. EuroIntervention. 2016 Nov 20;12(10):1298-1304. doi: 10.4244/EIJV12I10A213. PMID 27866140
- [Result] Hein-Rothweiler R, Jochheim D, Rizas K, Egger A, Theiss H, Bauer A, Massberg S, Mehilli J. Aortic annulus to left coronary distance as a predictor for persistent left bundle branch block after TAVI. Catheter Cardiovasc Interv. 2017 Mar 1;89(4):E162-E168. doi: 10.1002/ccd.26503. Epub 2016 Apr 1. PMID 27038099
- [Result] Jochheim D, Zadrozny M, Theiss H, Baquet M, Maimer-Rodrigues F, Bauer A, Lange P, Greif M, Kupatt C, Hausleiter J, Hagl C, Massberg S, Mehilli J. Aortic regurgitation with second versus third-generation balloon-expandable prostheses in patients undergoing transcatheter aortic valve implantation. EuroIntervention. 2015 Jun;11(2):214-20. doi: 10.4244/EIJV11I2A40. PMID 26093840
- [Result] Jochheim D, Abdel-Wahab M, Mehilli J, Ellert J, Wubken-Kleinfeld N, El-Mawardy M, Pache J, Massberg S, Kastrati A, Richardt G. Significant aortic regurgitation after transfemoral aortic valve implantation: patients' gender as independent risk factor. Minerva Cardioangiol. 2015 Oct;63(5):371-9. Epub 2015 Mar 27. PMID 25812583
- [Result] Jochheim D, Schneider VS, Schwarz F, Kupatt C, Lange P, Reiser M, Massberg S, Gutierrez-Chico JL, Mehilli J, Becker HC. Contrast-induced acute kidney injury after computed tomography prior to transcatheter aortic valve implantation. Clin Radiol. 2014 Oct;69(10):1034-8. doi: 10.1016/j.crad.2014.05.106. Epub 2014 Jul 10. PMID 25017451